CLINICAL TRIAL: NCT01434940
Title: Early Oculomotor Markers in Alzheimer's Disease: Test of Predictive Value in the Differential Diagnosis Depression/Alzheimer
Brief Title: Eye Movement Recording as an Early Differential Diagnostic Tool for Alzheimer/Depression
Acronym: MOMAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Laboratoire de psychologie EA 3188 (Unknown); Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier de Novillars (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N/2009/55
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer Disease; Depression
Keywords: Alzheimer disease; Depression; Differential diagnosis; Eye movement
MeSH Terms: conditions — Alzheimer Disease; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alzheimer (Experimental): Patients suffering of Alzheimer disease
  Interventions: Other: Eye movements will be recorded using video-oculography techniques based on both the corneal reflection principle and an infra-red light beam
- Depression (Experimental): Patients suffering from depression
  Interventions: Other: Eye movements will be recorded using video-oculography techniques based on both the corneal reflection principle and an infra-red light beam
- Healthy (Experimental): Healthy volunteers
  Interventions: Other: Eye movements will be recorded using video-oculography techniques based on both the corneal reflection principle and an infra-red light beam

INTERVENTIONS:
Other: Eye movements will be recorded using video-oculography techniques based on both the corneal reflection principle and an infra-red light beam — . The system named H6-HSCN by Applied Science Laboratories (ASL®) helps keep the patient's head fixed on a support, important for the elderly population. This system allows to capture data with good temporal resolution (sampling at 360Hz) and good spatial resolution (accuracy of 0.1° of visual angle) at a distance of about 70 cm from the screen test with a visual angle of 32.6°. Results will be processed with ASL Result Software.

SUMMARY:
The global aim of our study is to validate eye movement recording as an early differential diagnostic tool, in order to discriminate as early as possible between neurodegenerative dementias of Alzheimer type and depressive pseudodementias (DPD). The investigators want to put forward idiosyncratic oculomotor characteristics of Alzheimer's disease (AD) and DPD respectively. Eye movements are sensitive markers of neurological diseases and can be used in a variety of clinical neurological syndromes.

This study compares 3 groups of 98 patients: patients suffering of AD and DPD and healthy persons. The patients AD will be recruited in the Memory Centre of Resources and Research of Besançon and patients DPD will be selected in the psychiatric department of the University Hospital of Besançon. The control participants will be recruited from the entourage of researchers and patients. The selection of participants in the 3 different groups is based on clinical examinations in psychiatry and neurology and neuropsychological assessments. After giving informed consent, patients will be evaluated by a psychiatrist and a neuropsychologist. The complete assessment takes 150 minutes.

After having set up patients, eye movements will be recorded using video-oculography techniques. The following tasks are performed: the basic dynamic eye movements (latency, hypometric and hypermetric saccades, reaction time, saccade speed, accuracy, pupil diameter) will be evaluated by the pro-saccade, anti-saccade and predictive saccade tasks. The emotional connotation tasks will be assessed by scan of images pair with emotional connotation and portrait analysis. The assessment takes 30 minutes.

This study will include 3 groups:

* an Alzheimer group;
* a depressed group;
* a control group with healthy persons. The population of this study will be comprised of patients over age 60 with a visual acuity over 9/10, not diagnosed with eye disease and not neuropsychological sequelae that could disrupt the functioning oculomotor.

These people will be recruited on a voluntary basis, after notification and consent in the research center, the Psychiatry Clinical Department of the University Hospital of Besançon. This study was conducted over a period of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* subject whose visual acuity > 9/10
* subject without a diagnosis of eye disease
* subject without a neuropsychological sequelae
* for depressed patients :subject with a diagnosis of depression confirmed by a psychiatric evaluation and MADRS (Montgomery and Asberg Depression Rating Scale) score >25 and without cognitive impairment or any other psychiatric pathology and MMSE (Mini Mental State Examination)≥18 and without symptoms of AD
* for Alzheimer patients :subject with AD diagnosed according to NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke -Alzheimer's Disease and Related Disorders Association) criteria and MMSE ≥18 and without psychiatric disorder and MADRS score < 25
* for control patients : subject without AD, depression or any other psychiatric condition identified by the diagnostic criteria or cognitive disorders and MADRS score <25 and MMSE > 20

Exclusion Criteria:

* subject age under 60

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2010-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
pro-saccade task | session1: after psychiatric and neuropsychologic assessment
  The score differences to pro-saccade task between the 3 groups constitute the major research outcome measure used to measure the basic dynamic eye movements.
anti-saccade task | session 2: after session 1 (pro-saccade task)
  The score differences to anti-saccade task between the 3 groups consitute one of the major research outcome measure used to measure the basic dynamic eye movements.
predictive saccade task | session 3: after session 2 (anti-saccade task)
  The score differences to predictive saccade tasks between the 3 groups constitute one of the major research outcome measure used to measure the basic dynamic eye movements
scan of images pair with emotional connotation | session 4 : after session 3 (predictive saccade task)
  The score differences of scan of images pair with emotional connotation were used to evaluate the emotional tasks
portrait analysis | session 5: after session 4 (scan of images pair with emotional connotation)
  The score differences of portrait analysis were used to evaluate the emotional tasks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre VANDEL, Prof, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Univserity Hospital of Besançon - Psychiatry Department, Besançon, France